CLINICAL TRIAL: NCT07387068
Title: First-in-human, Open-label, Phase 1 Trial to Evaluate the Safety and Preliminary Efficacy of GEN1079 in Participants With Select Advanced Malignant Solid Tumors
Brief Title: Trial to Evaluate the Safety and Preliminary Efficacy of GEN1079 in Participants With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1079-01; 2025-523931-21 (Other: EU CT Number)
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Masking Description: In the dose escalation part (Part 1), participants will not be randomized. If more than 1 dose level (DL) is explored in the dose refinement part (Part 2) and Expansion (Part 3), participants will be randomized across the selected DLs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: GEN1079 Dose Escalation (Experimental): Cohorts of participants will receive escalating doses of GEN1079 in up to 5 DLs.
  Interventions: Drug: GEN1079
- Part 2: GEN1079 Dose Refinement (Experimental): Cohorts of participants will receive up to 3 DLs of based on data from the Dose Escalation.
  Interventions: Drug: GEN1079
- Part 3: Expansion (Experimental): Cohorts of participants will receive up to 2 DLs of GEN1079 based on data from Dose Escalation/Dose Refinement.
  Interventions: Drug: GEN1079

INTERVENTIONS:
Drug: GEN1079 — Concentrate for solution.

SUMMARY:
The purpose of this trial is to learn about the safety and effectiveness of the antibody GEN1079 in participants with certain types of cancer.

The trial has multiple parts. The first part of the trial tests different doses of GEN1079 to find out if it is safe and determine what are the best doses to use. The second and third parts continue to test the safety of and whether GEN1079 works in additional participants with specific cancer types and at doses chosen based on results from the previous parts of the trial.

For each participant, the trial will last approximately 33 to 67 weeks but this may vary for each person. This includes up to 21 days for screening prior to receiving trial treatment, approximately 6 to 12 weeks of treatment (the duration of treatment may vary for each participant), and approximately 24 to 52 weeks of follow up after trial treatment ends (the duration of follow up may vary for each participant). During the screening, tumor tissue either collected prior to this trial or freshly collected during screening will be provided by all participants.

Participation in the trial will require visits to the site, with more frequent visits at the start of treatment and then less frequent visits afterwards. At site visits, there will be various tests (such as blood draws) and procedures (such as recording of heart activity, computed tomography [CT] scans) to monitor whether the treatment is safe and effective.

All participants will receive active drug; no one will be given placebo.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1, open-label, multinational, dose escalation and expansion trial in participants with advanced selected solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

All Parts:

* Must have histologically confirmed selected solid cancers.
* Have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. The measurable lesion(s) must be outside the field of prior radiation therapy unless there is documented progression in the lesion(s).
* Must provide formalin-fixed paraffin-embedded tumor tissue (aspirates and bone specimens are not acceptable), archival or fresh, collected after discontinuation of their most recent anticancer treatment and prior to the first administration of GEN1079. If an archival specimen is unavailable, a procedure for obtaining a fresh tumor biopsy must be performed, provided it is performed according to standard of care and is deemed safe by the investigator.
* Has acceptable laboratory test results prior to trial treatment administration, including platelet count >150×10^9/litre (L).

Parts 1 and 2:

* Have histologically confirmed selected solid cancers that are metastatic or unresectable.
* Prior protocol defined therapy is permitted, with no restrictions on the number of prior lines of therapy received or the time since the most recent therapy.

Part 3:

* Have histologically confirmed selected solid cancer that is metastatic or unresectable.
* Must have received a defined number of prior lines of a protocol defined regimen.

Key Exclusion Criteria:

* Has intercurrent illness or known history of any of the following that could affect compliance with the protocol or interpretation of the results, including but not limited to:

  * Autoimmune diseases, eg, systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), neuromyelitis optica (NMO), myasthenia gravis (MG), cold agglutinin disease (CAD), atypical hemolytic uremic syndrome (aHUS), immunoglobulin A (IgA) nephropathy, inflammatory bowel disease (IBD; Crohn's and ulcerative colitis).
  * Grade ≥3 allergic reactions to prior monoclonal antibody therapy.
  * Known history of interstitial lung disease (ILD) Grade ≥3 or prior or ongoing noninfectious pneumonitis with evidence of progressive fibrotic changes on baseline imaging, unless clinically and radiologically stable for ≥6 months with preserved pulmonary function (eg, diffusing capacity of the lungs for carbon monoxide [DLCO] ≥ 50% predicted).
  * Disorders associated with platelet function defects, decreased number of platelets (eg, splenomegaly, chronic liver disease or bleeding disorders such as hemophilia or Von Willebrand disease), or a known history or high risk of bleeding events requiring transfusions or hospitalizations.
* Treatment with any plasma-based therapy within 7 days prior to Cycle 1 Day 1.
* Any history of intracerebral arteriovenous malformation (shunts), cerebral aneurysm, spinal cord compression (from disease), carcinomatous meningitis, or stroke. Note: Transient ischemic attack >1 month prior to screening is allowed.
* Participants who, in the event of a medical complication during the trial treatment period, would be unable to temporarily discontinue and restart anticoagulant/antiplatelet therapy using appropriate bridging strategies (eg, low molecular weight heparin) in alignment with local standard of care.

Note: Other protocol-defined Inclusion and Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Part 1 Dose Escalation: Number of Participants with Dose-limiting Toxicities (DLTs) | 21 days
Part 1 Dose Escalation and Part 2 Dose Refinement: Number of Participants with Adverse Events (AEs) | Up to a maximum of approximately 67 weeks
Part 3 Expansion: Objective Response Rate (ORR) | Up to a maximum of approximately 67 months

SECONDARY OUTCOMES:
Part 1 Dose Escalation and Part 2 Dose Refinement: ORR | Up to a maximum of approximately 67 weeks
Part 1 Dose Escalation and Part 2 Dose Refinement: Disease Control Rate (DCR) | Up to a maximum of approximately 67 weeks
Part 1 Dose Escalation and Part 2 Dose Refinement: Duration Of Response (DOR) | Up to a maximum of approximately 67 weeks
Part 1 Dose Escalation and Part 2 Dose Refinement: Time to Response (TTR) | Up to a maximum of approximately 67 weeks
Part 1 Dose Escalation and Part 2 Dose Refinement: Maximum Concentration (Cmax) of GEN1079 | Up to a maximum of approximately 12 weeks
Part 1 Dose Escalation and Part 2 Dose Refinement: Time to Cmax (Tmax) of GEN1079 | Up to a maximum of approximately 12 weeks
Part 1 Dose Escalation and Part 2 Dose Refinement: Trough Concentration (Ctrough) of GEN1079 | Up to a maximum of approximately 12 weeks
Part 1 Dose Escalation and Part 2 Dose Refinement: Area Under the Concentration-time Curve from Time 0 to Last Quantifiable Sample (AUClast) of GEN1079 | Up to a maximum of approximately 12 weeks
Part 1 Dose Escalation and Part 2 Dose Refinement: Number of Participants with Anti-drug Antibodies (ADA) Against GEN1079 | Up to a maximum of approximately 12 weeks
Part 3 Expansion: DCR | Up to a maximum of approximately 67 weeks
Part 3 Expansion: DOR | Up to a maximum of approximately 67 weeks
Part 3 Expansion: TTR | Up to a maximum of approximately 67 weeks
Part 3 Expansion: Number of Participants with AEs | Up to a maximum of approximately 67 weeks
Part 3 Expansion: Cmax of GEN1079 | Up to a maximum of approximately 12 weeks
Part 3 Expansion: Tmax of GEN1079 | Up to a maximum of approximately 12 weeks
Part 3 Expansion: Ctrough of GEN1079 | Up to a maximum of approximately 12 weeks
Part 3 Expansion: AUClast of GEN1079 | Up to a maximum of approximately 12 weeks
Part 3 Expansion: Number of Participants with ADAs Against GEN1079 | Up to a maximum of approximately 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab

IPD SHARING:
Plan to Share IPD: No